CLINICAL TRIAL: NCT04129879
Title: ABC Technique as a Novel Approach for Endometriosis Surgery
Brief Title: a Novel Surgical Approach for Endometriosis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AcibademU abc
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Endometriosis; Laparoscopy
Keywords: endometriosis; methylene blue dye
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: patients undergone for laparoscopic surgery for endometriosis had both approaches with either bare eye and with the help of methylene blue contrast agent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): all patients treated by conventional bare eye technique and then the use of methylene blue contrast technique to visualize endometriotic lesions perioperatively
  Interventions: Procedure: ABC technique

INTERVENTIONS:
Procedure: ABC technique — The intraperitoneal use of methylene blue diluted isotonic sodium chloride solution to visualize endometriotic lesions

SUMMARY:
Endometriosis is a chronic disease defined as the existence of endometrium like lesions outside of the uterine cavity. The diagnosis is based on examination of lesions under the microscope and capturing endometrial gland and stroma. The mostly used surgical technique to diagnose and treat endometriosis is laparoscopic surgery. In our novel technique for endometriosis surgery, we used methylene blue for its natural blue color to make endometriotic lesions more visible and to filter red, yellow and white colors reflecting from the peritoneal surface.

DETAILED DESCRIPTION:
Endometriosis is a chronic disease defined as existence of endometrium like lesions outside of the uterine cavity. The diagnosis is based on examination of lesions under microscope and capturing endometrial gland and stroma. The prevalence of endometriosis upon women on their reproductive ages, all over the world is at least 10%. This prevalence depends on surgically proven lesions that are excised, according to the this the real prevalence is still unknown because of underdiagnosis and being unable to capture endometriotic lesions.

Endometriosis is usually described as having three subtypes, which are peritoneal, ovarian endometriomas and deep infiltrative endometriosis (DIE). Peritoneal endometriosis is the most undiagnosed type according to lack of diagnostic tests and being unrecognizable on imaging modalities while ovarian endometriomas and deep infiltrative endometriosis lesions can be realized by ultrasound or MRI imaging. Also, these three subtypes are mostly existing together and even with uterine endometriosis which is named as adenomyosis. Considering the difficulties of capturing an endometriotic lesion most of the surgeries done for deep endometriosis or ovarian endometriomas usually fail upon insufficient excision of the disease.

The main presentations of endometriosis are pain and infertility. Whether it can be thought the most devastating anatomical lesion may cause more pain, the pain of endometriosis is usually unrelated with the characteristics of pathology or severity of the disease. Therefore, a small lesion even not visible to the naked eye may cause more pain than a large DIE nodule. This knowledge arises the importance of threating all lesions on a symptomatic patient with pain.

The mostly used surgical technique to diagnose and treat endometriosis is laparoscopic surgery. Under laparoscopic scope endometriotic lesions can bee seen in black, red, white colors and as flat or polypoid. Human eye can see wave lengths between 400-700 nm. And it is not always easy to visualize all pathologies even with the 4 to 40 times magnification of usual laparoscopic scopes. Human vision under white-light reflection cannot easily discriminate different tissue types. Making color contrasts make objects easy to be catch by human eye.

In our novel technique for endometriosis surgery we used methylene blue for its natural blue color to make endometriotic lesions more visible and to filter red, yellow and white colors reflecting from peritoneal surface.

ELIGIBILITY:
Inclusion Criteria:

* patients who have endometriosis
* patients who approved their data to be used for research manner
* operations with only peritoneal endometriosis

Exclusion Criteria:

* operations without the diagnosis of endometriosis
* patients who have not approved their data to be used for research manner
* operations which also include endometriomas and/or deep infiltrative endometriosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — it is a gynecologic situation
Enrollment: 115 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
number of samples taken from each region | retrospective 1 year period

SECONDARY OUTCOMES:
number of endometriosis positivity came out of each excision | retrospective 1 year period

CONTACTS AND LOCATIONS:
Locations (1):
- Bahar Yuksel, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Abesadze E, Sehouli J, Mechsner S, Chiantera V. Possible Role of the Posterior Compartment Peritonectomy, as a Part of the Complex Surgery, Regarding Recurrence Rate, Improvement of Symptoms and Fertility Rate in Patients with Endometriosis, Long-Term Follow-Up. J Minim Invasive Gynecol. 2020 Jul-Aug;27(5):1103-1111. doi: 10.1016/j.jmig.2019.08.019. Epub 2019 Aug 23. PMID 31449906